CLINICAL TRIAL: NCT05435755
Title: The Precise Transplantation of Human Amniotic Epithelial Stem Cells Into the Ventricle Through Surgical Robot in the Treatment of Parkinson's Disease.
Brief Title: Precise Transplantation of hAESCs Into the Ventricle for Parkinson's Disease.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020YFA0112600
Record Dates: First submitted 2022-03-15; First posted 2022-06-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; stem cell
MeSH Terms: conditions — Parkinson Disease | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study plans to recruit 12 patients who meet the criteria. 50 millions hAESCs will be transplanted to participants with PD.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hAESCs treatment (Experimental): A total of 6 times hAESCs transplants will be performed. 50 million (in 2ml) hAESCs will be transplanted into the ventricle of participants through the Ommaya sac (set as day 0 at the beginning of the trial). Subsequently, hAESCs ventricle transplants will be performed at 1 month ±5 days, 2 months ±5 days, 3 months ±5 days, 6 months ±5 days, and 9 months ±5 days after the first cell transplantation, with a volume of 50 million cells (in 2 ml) each time.
  Interventions: Biological: hAESCs treatment
- Control group (Placebo Comparator): Four times hAESCs transplants and two times placebo (cell preservation solution) injections will be performed by Ommaya sac. 50 million (in 2ml) hAESCs will be transplanted into the ventricle of participants (set as day 0 at the beginning of the trial). Subsequently, hAESCs will be transplanted into the ventricle for 3 times, respectively, at 1 month ±5 days , 2 months±5 days , and 3 months ±5 days after the first cell transplantation, with a volume of 50 million cells (in 2 ml) each time. Ventricle injection of 2 ml placebo (cell preservation solution) will be performed at 6 months ±5 days and 9 months ±5 days after the first cell transplantation.
  Interventions: Biological: placebo (saline)

INTERVENTIONS:
Biological: hAESCs treatment — Precise Transplantation of hAESCs Into the Ventricle for Parkinson's Disease.
  Arms: hAESCs treatment
Biological: placebo (saline) — 2 times placebo (normal saline) injections as control group
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the safety of multiple treatments of hAESCs treatments, while exploring the effectiveness of hAESCs treatments for PD.

DETAILED DESCRIPTION:
The study plans to use randomized controlled trial and recruit 12 participants with Idiopathic Parkinson's disease. The trial will be divided into two groups, hAESCs treatment group and control group, each group 6 subjects. Through surgical robot technology, hAESCs will be precisely multiple transplanted into the lateral ventricles, that is two times consolidation hAESCs treatments or placebo were added to the four times basic hAESCs treatments. Therapeutic safety and effectiveness of multiple treatments of hAESCs on PD will be evaluated to further develop the optimal stem cell treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. 30-70 years old, with more than 5 years primary Parkinson's disease history, male or female;
2. The "off-age" UPDRS exercise score is between 38 and 70 points, two times before the operation, the "down period" UPDRS exercise score was stable, that is, (high value - low value) / high value ≤ 10%;
3. The Parkinson treatment is stable for more than 3 months;
4. Levodopa treatment was effective;
5. No general anesthesia contraindications, no contraindications to stereotactic surgery and other conditions that interfere with clinical evaluation;
6. No abnormalities affecting cell transplantation were found through the cranial MRI;
7. Patients shall be properly cared during treatment, and caregivers can provide transplantation situations and assistance to the researcher if necessary.

Exclusion Criteria:

1. Atypical Parkinson's disease, such as Parkinson's syndrome, secondary Parkinson's disease;
2. Only having tremor syndrome;
3. "off period" or "on period" has serious movement disorders and cannot complete any routine exercise tasks;
4. Symptoms of severe neurological deficits caused by other diseases;
5. Severe mental symptoms or dementia;
6. Patients are unwilling to cooperate or incapable of completing self-evaluation, and cannot complete the evaluator with the help of a doctor;
7. History of striatum or extrapyramidal surgery, including deep brain stimulation (DBS);
8. Injecting apomorphine treatment;
9. Abnormal blood coagulation or ongoing anticoagulation therapy;
10. Women of childbearing age who do not take effective contraception;
11. Pregnant or lactation;
12. Patients who have participated in other clinical studies of drugs or medical devices within 3 months;
13. Botox toxin, phenol, subarachnoid injection of baclofen or interventional therapy for the treatment of dystonia or spasticity within 6 months;
14. History of seizures or prophylactic anti-epileptic drugs;
15. Alcohol or drug abuse;
16. Severe cognitive impairment, depression, or behavioral disorder, defined as the Mini-Mental State Assessment Scale (MMSE) of less than 26 points, and the Hamilton Depression Rating Scale (HAMD) of greater than 35 points;
17. Malignant tumor or active infection within 5 years;
18. Serum virology showed positive results for hepatitis C virus (HCV) , treponema pallidum (TP) or HIV; Active hepatitis B (hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) positive, and peripheral blood HBV DNA titer ≥1×10^3 IU/ mL);
19. Abnormal liver and kidney function tests in the laboratory, liver and kidney function is defined as Alanine aminotransferase（ALT), Aspartate aminotransferase（AST) is less than 2.5 times the upper limit of normal, blood urea nitrogen (BUN) and Creatinine（Cr) are less than the upper limit of normal.
20. Other conditions considered ineligible for inclusion by the investigator.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-02 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse event (AE), serious adverse event(SAE) and adverse events of special interest(AESI) | 12 Months
  AE occurring throughout the study period will be evaluated using the CTCAE V5.0 standard. AE/SAE and AESI were evaluated after Ommaya sac installation by laboratory examination, measurement of vital signs, physical examination, and subjects' symptoms to detect new abnormalities and/or deterioration of previous conditions and evaluate the safety of the study.
  AESI is defined as intracranial infection, hemorrhage, rejection, and edema within 7 days after Ommaya sac installation, as well as acute allergic reactions and ectopic mass formation associated with study therapy.

SECONDARY OUTCOMES:
Changes in Unified Parkinson's Disease Rating Scale (UPDRS) in OFF state between the experimental group and the control group at 12 months after the first hAESCs treatment | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  UPDRS is used for evaluating the impairment and disability associated with Parkinson's Disease (PD). It consists of four sections: (1) Mentation, behavior, and mood; (2) Activities of daily living (ADLs); (3) Motor; and (4) Complications.
  The UPDRS score ranges from 0 to 199, with higher score indicating greater disability
Changes in the Hoehn and Yahr scale | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  Hoehn and Yahr scale is used to provide a general estimate of clinical function of PD patients, combining functional deficits (disability) and objective signs (impairment). The Hoehn and Yahr score ranges from 0 to 5, with higher score indicating higher dysfunction of PD patients.
Changes in the Schwab and England score | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  The Schwab and England score develop a scale that describes the capacity of daily living shown by a PD patients. It measures the following three areas: dependence, abilities, and awareness. The Schwab and England score range from o% to 100%, with higher scores indicating greater healthy status.
Changes in the Parkinson's Disease Questionnaire (PDQ-39) | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  PDQ-39 provides the evidence of the quality of life of a PD patient. The higher the score, the lower the quality of life of PD patients.
Changes in the Hamilton Depression (HAMD) Scale | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  HAMD is the most widely used scale in clinical evaluation of depression in PD patients. This project takes 8 points as the critical value of depression, and the total score over 35 points is considered as severe depression, more than 20 points is likely to be diagnosed with depression, less than 8 points is not depressed.
Differences in biochemical indicators of cerebrospinal fluid | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  Cerebrospinal fluid indicator tests include biochemical indicators and the following parameters: Dopamine (DA), high vanillic acid (HVA), 5-hydroxytryptamine (5-HT), 5-hydroxyindoleacetic acid (5-HIAA), norepinephrine (MHPG), α synuclein (α-synuclein), amyloid deposition (Aβ42), Tau protein (Tau) Protein, Neurofilament light (NF-L), and yKL-40 (YKL-40).
Cranial dopamin transporter measured by positron emission tomography (PET)- magnetic resonance imaging (MRI) | 4 month, 6 month, 12 month
  Changes of cranial expression of dopamine transporter investigated by PET-MR
Glucose metabolism measured by 18F-Fluoro-2-deoxy-glucose (FDG) PET scan | 4 month, 6 month, 12 month
  Changes of cranial glucose metabolism investigated by PET-MR

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Wu, Dr, Principal Investigator — Shanghai East Hospital, China
Locations (1):
- Jingwen Wu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No